CLINICAL TRIAL: NCT00297570
Title: Imatinib Versus Imatinib and Peg-Interferon in Patients With Ph+ CML and Complete Cytogenetic Response After Imatinib Therapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-06-4015-IH-CTIL
Record Dates: First submitted 2006-02-27; First posted 2006-02-28 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Leukemia, Myeloid, Philadelphia-Positive
Keywords: CML; Imatinib; Pegylated Interferon; Philadelphia Positive CML
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Pegylated Interferon and Imatinib

SUMMARY:
The study is controlled and randomized in Philadelphia-positive chronic myeloid leukemia (Ph+ CML) patients with complete cytogenetic response after more than one year of imatinib therapy. The aim is to explore a possible benefit in the addition of peg-interferon (Peg-IFN) to imatinib, in terms of the rate of achievement, molecular remission, and response duration.

ELIGIBILITY:
Inclusion Criteria:

* Ph+ CML patients in complete cytogenetic response (CCR) after more than 1 year of imatinib therapy.

Exclusion Criteria:

* Patients in imatinib study
* Patients with a history of intolerability to interferon.
* Patients with less than CCR or less than one year of imatinib therapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-02

CONTACTS AND LOCATIONS:
Overall Officials: Izhar Hardan, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Department of Hematology, Sheba Medical Center, Tel Litwinsky, Tel-Hashomer, Israel

REFERENCES:
- [Derived] Hardan I, Stanevsky A, Volchek Y, Tohami T, Amariglio N, Trakhtenbrot L, Koren-Michowitz M, Shimoni A, Nagler A. Treatment with interferon alpha prior to discontinuation of imatinib in patients with chronic myeloid leukemia. Cytokine. 2012 Feb;57(2):290-3. doi: 10.1016/j.cyto.2011.11.018. Epub 2011 Dec 13. PMID 22169779